CLINICAL TRIAL: NCT04814836
Title: Clinical Evaluation of Cervical Composite Restorations Placed Using Universal Adhesive in Different Modes and Different Etching Methods
Brief Title: Laser Etching Effect on Application Mode of Universal Adhesive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, A Ruya Yazici, Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA180076
Record Dates: First submitted 2021-03-11; First posted 2021-03-24 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy Participant
Keywords: non-carious cervical lesions; universal adhesives; laser etching
MeSH Terms: interventions — phosphoric acid

STUDY DESIGN:
Intervention Model Description: This study was carried out to investigate different etching methods used for application modes of universal adhesive on clinical performance of non-carious cervical lesions. The 35% phosphoric acid (K-ETCHANT) or Er,Cr:YSGG laser (2780 nm, Waterlase MD, BioLase Technology, Inc.) etching was applied to the tooth before these application modes in order to bond the universal adhesive, Clearfil Universal Bond Quick. Accordingly, the restorations were completed with 5 different application methods to five different teeth. The allocation of etching method and application mode on each tooth was determined in an order that was assigned by Biostatistics Department. This randomization was blinded to participants and evaluators. It was not known which etching method and application mode was applied to which teeth of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group I (Other): Total-etch mode with 35% phosphoric acid
  Interventions: Procedure: Total-etch mode with 35% phosphoric acid (K-ETCHANT) (TE-A group)
- Group II (Other): Selective-etch mode with 35% phosphoric acid
  Interventions: Procedure: Selective-etch mode with 35% phosphoric acid (K-ETCHANT) (SE-A group)
- Group III (Other): Total-etch mode with laser (Er,Cr:YSGG)
  Interventions: Procedure: Total-etch mode with Er, Cr: YSGG laser (Waterlase MD) (TE-L group)
- Group IV (Other): Selective-etch mode with laser (Er,Cr:YSGG)
  Interventions: Procedure: Selective-etch mode with Er, Cr: YSGG laser (Waterlase MD) (SE-L group).
- Group V (Other): Self-etch mode
  Interventions: Procedure: Self-etch mode Clearfil Universal Bond Quick (Kuraray, Japan) (SE group)

INTERVENTIONS:
Procedure: Total-etch mode with 35% phosphoric acid (K-ETCHANT) (TE-A group) — 35% phosphoric acid was applied to enamel and dentin for 10 s, washed and dried for 5 s. The universal adhesive, Clearfil Universal Bond Quick (CBQ) was applied to enamel and dentin surfaces with a single-use applicator, then gently air-dried for 5 s without waiting, and light-cured for 10 s.
  Arms: Group I
Procedure: Selective-etch mode with 35% phosphoric acid (K-ETCHANT) (SE-A group) — 35% phosphoric acid was used only on enamel for 10 s, then washed and dried for 5 seconds. Subsequently, the adhesive was applied in a similar manner to the TE-A group.
  Arms: Group II
Procedure: Total-etch mode with Er, Cr: YSGG laser (Waterlase MD) (TE-L group) — the enamel margin and dentin surfaces of lesions were irradiated with an Er,Cr:YSGG laser (2780 nm, Waterlase MD, BioLase Technology, Inc., San Clemente, CA). Then the adhesive was applied in a similar manner to the TE-A group.
  Arms: Group III
Procedure: Selective-etch mode with Er, Cr: YSGG laser (Waterlase MD) (SE-L group). — The laser system was applied in the same way as described in the TE-L group only on enamel surface. Subsequently, the adhesive was applied in the same way as described in the TE-A group.
  Arms: Group IV
Procedure: Self-etch mode Clearfil Universal Bond Quick (Kuraray, Japan) (SE group) — Universal adhesive system (CBQ) was applied to enamel and dentin surfaces without any previous etching. Then gently air-dried for 5 s without waiting, and light-cured for 10 s.
  Arms: Group V

SUMMARY:
To evaluate the clinical performance of the restorations by applying the universal adhesive in different modes under the influence of different surface treatments, with Erbium Chromium:Yttrium-Scandium-Gallium-Garnet (Er,Cr:YSGG) laser and acid etching in non-carious cervical lesions.

DETAILED DESCRIPTION:
Forty-one patients (at least five non-carious cervical lesions) have participated in this study. The non-carious cervical lesions in each patient were divided into five groups (total-etch mode with phosphoric acid, selective-etch mode with phosphoric acid, total-etch mode with laser, selective-etch mode with laser and self-etch mode) according to different modes and application methods of universal adhesive (Clearfil Universal Bond Quick, Kuraray). Lesions were restored with a resin composite, Clearfil Majesty ES-2 (Kuraray). All restorative procedures were performed by a single operator. Restorations were evaluated at one week (baseline), at 6-, 12-, 18- and 24-month according to modified USPHS criteria (retention, marginal discoloration, marginal adaptation, color match, postoperative sensitivity, and secondary caries) by two experienced and calibrated investigators.

ELIGIBILITY:
Inclusion Criteria:

* Participants were 18 years of age or older,
* no possible health problems (such as allergies) related to resin-based restorations,
* good general health,
* having at least five non-carious cervical lesions.
* The depth of the lesions were at least 1 mm, without carious, not previously restored, having teeth with vital, enamel and dentin tissue.

Exclusion Criteria

* Participant had fewer than 20 teeth,
* having poor oral hygiene,
* uncontrolled periodontal disease,
* xerostomia,
* pregnancy or breastfeeding possible health problems (such as allergy) related to resin-based restorations,
* having bleaching treatment or orthodontic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Retention, | From baseline to 2 year the change of restorations was evaluated
  The retention criterion determines how long a restorative material functions in the oral environment, it is the most important criterion that shows the success of the material.
  Alpha: The restoration is present. Charlie: The restoration is absent.
Marginal Discoloration | From baseline to 2 year the change of restorations was evaluated
  The marginal discoloration that occur at the edge staining restoration boundaries are generally thought to be due to microleakage.
  Alpha: No discoloration at margins. Bravo: Shallow discoloration, clinically acceptable. Charlie: Deep discoloration clinically unacceptable.
Marginal Adaptation | From baseline to 2 year the change of restorations was evaluated
  Marginal adaptation is achieved by fully ensuring the integrity of the tooth-restoration joint border.
  Alpha: Restoration is closely adapted to the tooth. Bravo: Visible evidence of a crevice along the margin, dentin not exposed, clinically acceptable.
  Charlie: Explorer penetrates into crevice, dentin is exposed; clinically unacceptable.
Color match | From baseline to 2 year the change of restorations was evaluated
  Color match is the evaluation of the restoration according to the darkening or lightening of the color, taking into account the tooth tissue surrounding restoration.
  Alpha:Matches tooth. Bravo: Acceptable mismatch. Charlie:Unacceptable mismatch.
Post-op Hypersensitivity | From baseline to 2 year the change of restorations was evaluated
  Determination of sensitivity after restorations are placed. Alpha: Absent. Charlie: Present; clinically unacceptable.
Secondary Caries | From baseline to 2 year the change of restorations was evaluated
  Secondary caries is the progression of caries in the tooth tissue adjacent to the restorations. Caries formation means restoration failure.
  Alpha: Absent. Charlie: Present; clinically unacceptable.

CONTACTS AND LOCATIONS:
Overall Officials: A. Ruya Yazici, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Atalay C, Uslu A, Yazici AR. Does laser etching have an effect on application mode of a universal adhesive?-A microleakage and scanning electron microscopy evaluation. Microsc Res Tech. 2021 Jan;84(1):125-132. doi: 10.1002/jemt.23573. Epub 2020 Aug 27. PMID 32852126
- [Background] Atalay C, Ozgunaltay G, Yazici AR. Thirty-six-month clinical evaluation of different adhesive strategies of a universal adhesive. Clin Oral Investig. 2020 Apr;24(4):1569-1578. doi: 10.1007/s00784-019-03052-2. Epub 2019 Aug 30. PMID 31468262
- See also: Related Info — https://link.springer.com/article/10.1007/s00784-019-03052-2